CLINICAL TRIAL: NCT05038800
Title: A Phase 1b Study to Evaluate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics of MK-0482 in Participants With Relapsed or Refractory Acute Myeloid Leukemia or Chronic Myelomonocytic Leukemia
Brief Title: A Study to Evaluate MK-0482 for Relapsed/Refractory Acute Myeloid Leukemia (AML) or Chronic Myelomonocytic Leukemia (CMML) (MK-0482-002)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0482-002; MK-0482-002 (Other: MSD); 2023-003740-27-00 (Registry Identifier: EU CT); U1111-1287-5269 (Registry Identifier: UTN); 2022-003740-27 (EudraCT Number)
Record Dates: First submitted 2021-08-24; First posted 2021-09-09 (Actual); Results first posted 2024-12-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia; Relapsed or Refractory Chronic Myelomonocytic Leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- MK-0482 7.5 mg Q3W (Experimental): Participants will receive 7.5 mg of MK-0482 via intravenous (IV) infusion on Day 1 of each 21-day cycle (every 3 weeks [Q3W]) for up to 35 cycles (approximately 24 months).
  Interventions: Biological: MK-0482
- MK-0482 25 mg Q3W (Experimental): Participants will receive 25 mg of MK-0482 via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 24 months).
  Interventions: Biological: MK-0482
- MK-0482 75 mg Q3W (Experimental): Participants will receive 75 mg of MK-0482 via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 24 months).
  Interventions: Biological: MK-0482
- MK-0482 225 mg Q3W (Experimental): Participants will receive 225 mg of MK-0482 via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 24 months).
  Interventions: Biological: MK-0482
- MK-0482 750 mg Q3W (Experimental): Participants will receive 750 mg of MK-0482 via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 24 months).
  Interventions: Biological: MK-0482

INTERVENTIONS:
Biological: MK-0482 — IV infusion

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and recommended Phase 2 dose (RP2D) of MK-0482. There are 2 parts of this study. Part 1 is a dose escalation which will follow an accelerated titration design (ATD) for participants with relapsed/refractory (R/R) AML or CMML. Part 2 is a dose expansion for participants with R/R AML.

DETAILED DESCRIPTION:
In Part 1, single participants will be enrolled sequentially into escalating dose levels. Progression from one dose level to the next higher dose level will be based on the evaluation of dose-limiting toxicity (DLT). Once a preliminary RP2D is identified in Part 1, approximately 10 to 15 additional participants with R/R AML will be enrolled at the RP2D for Part 2.

ELIGIBILITY:
Inclusion Criteria:

-Has confirmed diagnosis of AML with myelomonocytic or monoblastic/monocytic differentiation per World Health Organization (WHO) 2016 criteria and with confirmed refractory or relapsed disease (i.e., ≥5% blast in bone marrow or in peripheral blood) after treatment with available therapies known to benefit participant's AML subtypes or has a known diagnosis of CMML per WHO criteria [2017] with confirmed refractory or released disease after treatment with available therapies known to be active for CMML.

Exclusion Criteria:

* Has active central nervous system (CNS) leukemia.
* Has isolated extramedullary disease, i.e., no leukemic involvement in bone marrow or peripheral blood.
* Has diagnosis of acute promyelocytic leukemia or participants with known Philadelphia chromosome positive (Ph+) AML.
* Has received previous allogeneic stem cell transplant or organ transplant within 60 days of the start of study treatment.
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 1 year.
* Has a history of any of the following cardiovascular conditions within 6 months of screening: myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, coronary artery bypass graft, or pulmonary embolism; has New York Heart Association (NYHA) Class III or IV congestive heart failure.
* Has had a severe hypersensitivity reaction to treatment with a monoclonal antibody (mAB) and or any components of the study intervention, MK-0482.
* Has an active uncontrolled infection requiring directed therapy.
* Has immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, or disseminated intravascular coagulation.
* Has known human immunodeficiency virus (HIV) and/or hepatitis B or C infections, or is known to be positive for HBsAg/ Hepatitis B virus (HBV) Deoxyribonucleic acid (DNA) or hepatitis C antibody or Ribonucleic acid (RNA).
* Has known psychiatric or substance abuse disorders (verbally reported) that would interfere with the participant's ability to cooperate with the requirements of the study.
* Is pregnant or breast feeding or expecting to conceive or father children within the projected duration of the study, starting with the Screening Visit through 120 days after the last dose of study intervention.
* Has received systemic anticancer therapy, radiotherapy, or surgery within 2 weeks before the start of study treatment.
* Has received hematopoietic cytokines (Granulocyte Colony Stimulating Factor (G-CSF), Granulocyte Macrophage (GM)-CSF, or erythropoietin) within 2 weeks prior to start of study treatment.
* Has received a live or live attenuated vaccine within 30 days before the first dose of study medication.
* Is currently participating and receiving study intervention in a study of an investigational agent or has participated and received study intervention in a study of an investigational agent or has used an investigational device within 14 days of administration of MK-0482.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior the first dose of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (5):
- United States (2):
  - Roswell Park Cancer Institute ( Site 0006), Buffalo, New York
  - University of Texas MD Anderson Cancer Center ( Site 0004), Houston, Texas
- Israel (2):
  - Hadassah Medical Center ( Site 0100), Jerusalem
  - Sheba Medical Center-Hemato Oncology ( Site 0101), Ramat Gan
- Hospital Universitario de Salamanca - Complejo Asistencial U-Servicio de Hematologia ( Site 0301), Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26660&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirteen participants enrolled, of which 12 received study treatment in Part 1 of the study (dose-escalation).
  Part 2 of the study (dose expansion) was not conducted due to early termination of the study.
Groups:
- MK-0482 7.5 mg Q3W: Participants were to receive 7.5 mg of MK-0482 via intravenous (IV) infusion on Day 1 of each 21-day cycle (every 3 weeks [Q3W]) for up to 35 cycles (approximately 24 months).
- MK-0482 25 mg Q3W: Participants were to receive 25 mg of MK-0482 via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 24 months).
- MK-0482 75 mg Q3W: Participants were to receive 75 mg of MK-0482 via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 24 months).
- MK-0482 225 mg Q3W: Participants were to receive 225 mg of MK-0482 via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 24 months).
- MK-0482 750 mg Q3W: Participants were to receive 750 mg of MK-0482 via IV infusion on Day 1 of each 21-day cycle (Q3W) for up to 35 cycles (approximately 24 months).
Period: Overall Study
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Started | 1 | 1 | 5 | 3 | 3
Treated | 1 | 1 | 5 | 3 | 2
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 5 | 3 | 3
Not completed — Death | 1 | 1 | 5 | 3 | 1
Not completed — Randomized By Mistake Without Study Treatment | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W | Total
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 3 | 13
Age, Customized [Number; unit: Participants]
  0 to 17 years | 0 | 0 | 0 | 0 | 0 | 0
  18 to 64 years | 0 | 0 | 2 | 1 | 0 | 3
  65 to 84 years | 1 | 1 | 3 | 2 | 3 | 10
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 1 | 1 | 4
  Male | 1 | 1 | 3 | 2 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants are indicated as "not reported" due to the risk of identification of a person.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 0 | 0 | 5 | 3 | 2 | 10
    Unknown or Not Reported | 1 | 1 | 0 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants are indicated as "not reported" due to the risk of identification of a person.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 1 | 0 | 1 | 2
    White | 0 | 0 | 4 | 3 | 2 | 9
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced a Dose-Limiting Toxicity (DLT)
Description: DLTs were defined as any of the following assessed as treatment-related by investigator (with pre-specified exceptions): Grade (Gr) 4 non-hematologic toxicity; Gr 3 non-hematologic toxicity; Gr 3 or Gr 4 non-hematologic laboratory value if: clinically significant medical intervention was required to treat the participant, the abnormality led to hospitalization, the abnormality persisted for >1 week, electrolyte imbalances that lasted >48 hours despite optimal therapy, or the abnormality resulted in a drug-induced liver injury; Gr 4 neutropenia and/or thrombocytopenia lasting >14 days; >2 week-delay in starting Cycle 2 due to treatment-related toxicity; treatment-related toxicity resulting in treatment discontinuation during DLT evaluation period; missing >25% of MK-0482 dose during DLT evaluation period resulting from treatment-related adverse event (AE); or Gr 5 toxicity. The percentage of participants that experienced a DLT was reported for each arm.
Time Frame: Cycle 1 (up to 21 days)
Population: The DLT evaluable population included all allocated participants in Part 1 (dose escalation) who received at least 1 dose of study intervention and met the criteria for DLT evaluability (i.e finished Cycle 1 without a DLT, or experienced a DLT in Cycle 1).
Measure: Number (80% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 2
Percentage of Participants | 0.0 [0.0 to 55.3] | 0.0 [0.0 to 55.3] | 0.0 [0.0 to 23.5] | 0.0 [0.0 to 33.1] | 0.0 [0.0 to 41.5]

2. Primary Outcome: Number of Participants Who Experience at Least One Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced at least one AE was reported for each arm.
Time Frame: Up to approximately 10 months
Population: All allocated participants who received at least 1 dose of study intervention were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 2
Participants | 1 | 1 | 5 | 3 | 2

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinued study treatment due to an AE was reported for each arm.
Time Frame: Up to approximately 4 months
Population: All allocated participants who received at least 1 dose of study intervention were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 2
Participants | 0 | 0 | 1 | 0 | 0

4. Secondary Outcome: Maximum Concentration (Cmax) of MK-0482
Description: Cmax was defined as the maximum concentration of MK-0482 observed in plasma. Blood samples were collected pre-dose and post-dose at designated timepoints to determine Cmax of MK-0482.
Time Frame: Cycle 1: Pre-dose and Days 1, 2, 4, 8, and 15 post-dose. Cycle=21 days.
Population: All allocated participants who received at least 1 dose of study intervention, were compliant with the study procedures, and had available data from at least 1 treatment dose were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 2
ng/mL | 1490 (NA) — NA = Geometric coefficient of variation values were not reported when N < 2. | 5610 (NA) — NA = Geometric coefficient of variation values were not reported when N < 2. | 22000 (28.1) | 53400 (31.0) | 125000 (24.6)

5. Secondary Outcome: Minimum Concentration (Cmin) of MK-0482
Description: Cmin (or Ctrough) was defined as the lowest concentration of MK-0482 reached during a dosing interval (time interval between administration of two doses). Blood samples were collected pre-dose and post-dose at designated timepoints to determine Cmin of MK-0482.
Time Frame: Cycle 1: Pre-dose and Days 1, 2, 4, 8, and 15 post-dose. Cycle=21 days.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 2
ng/mL | 0.00 (NA) — NA = Geometric coefficient of variation values were not reported when N < 2. | 0.00 (NA) — NA = Geometric coefficient of variation values were not reported when N < 2. | 415 (2077.3) | 11200 (34.6) | 24500 (61.9)

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 21 Days (AUC0-21) of MK-0482
Description: AUC0-21 was defined as the area under the plasma concentration-time curve from time zero to 21 days. Blood samples were collected pre-dose and post-dose at designated timepoints to determine AUC0-21 of MK-0482.
Time Frame: Cycle 1: Pre-dose and Days 1, 2, 4, 8, and 15 post-dose. Cycle=21 days.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ng/mL
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 2
day*ng/mL | 3110 (NA) — NA = Geometric coefficient of variation values were not reported when N < 2. | 17200 (NA) — NA = Geometric coefficient of variation values were not reported when N < 2. | 105000 (64.5) | 521000 (22.9) | 885000 (12.4)

7. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-0482
Description: Tmax was defined as the time to maximum concentration of MK-0482 observed in plasma. Blood samples were collected pre-dose and post-dose at designated timepoints to determine Tmax of MK-0482.
Time Frame: Cycle 1: Pre-dose and Days 1, 2, 4, 8, and 15 post-dose. Cycle=21 days.
Population: as for outcome 4
Measure: Median (Full Range); unit: Days
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 2
Days | 0.04 [0.04 to 0.04] | 0.04 [0.04 to 0.04] | 0.04 [0.03 to 0.05] | 0.02 [0.02 to 0.03] | 0.03 [0.02 to 0.03]

8. Secondary Outcome: Plasma Elimination Terminal Half-life (t½) of MK-0482
Description: t½ was defined as the time required to divide the MK-0482 plasma concentration by two after reaching pseudo-equilibrium. Blood samples were collected pre-dose and post-dose at designated timepoints to determine t½ of MK-0482.
Time Frame: Cycle 1: Pre-dose and Days 1, 2, 4, 8, and 15 post-dose. Cycle=21 days.
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 2
Days | NA (NA) — NA = t½ and its corresponding geometric coefficient of variation were not calculated due to insufficient samples in the terminal phase to estimate lambda_z. | 2.46 (NA) — NA = Geometric coefficient of variation values were not reported when N < 2. | 3.69 (73.9) | 11.2 (34.7) | 11.2 (23.6)

9. Secondary Outcome: Complete Remission (CR) Rate
Description: CR Rate was assessed by the investigator per 2017 European Leukemia Net (ELN) Response Criteria for Acute Myeloid Leukemia (AML) and was defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count (ANC) ≥1.0 × 10^9/L (1000/µL); and platelet count ≥100 × 10^9/L (100,000/µL). The percentage of participants with CR (CR Rate) was reported for each arm.
Time Frame: Up to approximately 10 months
Population: All allocated participants who received at least 1 dose of study intervention and had a baseline assessment were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 1
Percentage of Participants | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 97.5]

10. Secondary Outcome: Composite CR Rate
Description: Composite CR rate was assessed by the investigator per 2017 ELN Response Criteria for AML and was defined as CR plus CR with incomplete recovery (CRi). CR was defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC ≥1.0 × 10^9/L (1000/µL); and platelet count ≥100 × 10^9/L (100,000/µL). CRi was defined as all CR criteria except for residual neutropenia (<1.0 × 10^9/L [1000/µL]) or thrombocytopenia (<100 × 10^9/L [100,000/µL]). The percentage of participants with Composite CR (Composite CR Rate) was reported for each arm.
Time Frame: Up to approximately 10 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 1
Percentage of Participants | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 97.5]

11. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was assessed by the investigator per 2017 ELN Response Criteria for AML and was defined as the combined percentage of participants with CR, CRi, and partial remission (PR). CR was defined as bone marrow blasts <5%; absence of circulating blasts and blasts with Auer rods; absence of extramedullary disease; ANC ≥1.0 × 10^9/L (1000/µL); platelet count ≥100 × 10^9/L (100,000/µL)]. CRi was defined as all CR criteria except for residual neutropenia (<1.0 × 10^9/L [1000/µL]) or thrombocytopenia (<100 × 10^9/L [100,000/µL]). PR was defined as all hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pre-treatment bone marrow blast percentage by at least 50%). ORR was reported for each arm.
Time Frame: Up to approximately 10 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
Number analyzed (Participants) | 1 | 1 | 5 | 3 | 1
Percentage of Participants | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 97.5]

ADVERSE EVENTS:
Time Frame: Up to approximately 10 months
Description: All-Cause Mortality was reported for all randomized participants.
  Serious AEs and Other AEs were reported for all randomized participants who received at least 1 dose of study treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | MK-0482 7.5 mg Q3W | MK-0482 25 mg Q3W | MK-0482 75 mg Q3W | MK-0482 225 mg Q3W | MK-0482 750 mg Q3W
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 5/5 | 3/3 | 1/3
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/5 | 2/3 | 2/2
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 4/5 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0482 7.5 mg Q3W (N=1) | MK-0482 25 mg Q3W (N=1) | MK-0482 75 mg Q3W (N=5) | MK-0482 225 mg Q3W (N=3) | MK-0482 750 mg Q3W (N=2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peri-implantitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0482 7.5 mg Q3W (N=1) | MK-0482 25 mg Q3W (N=1) | MK-0482 75 mg Q3W (N=5) | MK-0482 225 mg Q3W (N=3) | MK-0482 750 mg Q3W (N=2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papulosquamous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with ICMJE authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/00/NCT05038800/Prot_SAP_000.pdf